CLINICAL TRIAL: NCT03752346
Title: Effectiveness of Multimodal Exercise Program on Depression and Health-Related Quality of Life in Patients With Parkinson's Disease
Brief Title: Multimodal Exercise Program on Parkinson's Disease Patients With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 151223
Record Dates: First submitted 2018-10-31; First posted 2018-11-26 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-10

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; A Multimodal Exercise Program; Aerobic Exercise; Depression; Health Related Quality of Life
MeSH Terms: conditions — Parkinson Disease; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (No Intervention): Control group maintained their regular lifestyle and received the routine care
- exercise group (Experimental): Participants in the exercise group (EG) were instructed to engage performed exercise at least 3 times per week (30-50 minutes) or 10-15 minutes per section every day to accumulate 150 minutes per week for 8 weeks using disc (DVD) at home. Main exercise was moderate intensity aerobic exercise, an intensity of 55-70% of the heart rate reserve (HR max).
  Interventions: Other: exercise group

INTERVENTIONS:
Other: exercise group — A step aerobics exercise lasted a total 30 minutes, including:
  1. a warm-up with 10 minutes of stretching exercises.
  2. A step aerobics exercise (step aerobics for 30 minutes; step by step, step exercise, or stepping the ground repetitively)23,24 a total of 30 minutes then cool down (5 minutes).
  3. Resistance training (10 minutes), stretching and relaxation for 10-15 minutes.
  Arms: exercise group

SUMMARY:
Depression symptoms are common in Parkinson's Disease, it affects health-related quality of life. The evidence showed that exercise improved depression and HRQOL in PD patients. However, studies rarely considered the appropriate exercise program for PD patients, we want to find the best exercise program for PD patients.

DETAILED DESCRIPTION:
Objective: Evaluate the effectiveness of a 8-week multimodal exercise program on depression and HRQOL in PD Patients.

Methods: Single-blinded, randomized controlled trial, from March 2016 to January 2017. Ninety-eight patients recruited to 2 groups: exercise group (n = 49) and control group (n = 49). The primary outcomes were depression and HRQOL; the secondary outcomes were activity of daily living, motor ability, fatigue, sleep quality and anxiety. Data collection at baseline, week 4 and 8 after intervention. Intervention were Multimodal Exercise Program, at least three times (30 - 50 minutes per section) a week or 10-15 minutes per section every day to accumulate 150 minutes a week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* be diagnosed PD in Hoehn and Yahr stage I-II22
* under stable medication treatment at least 3 months
* no disease limiting the patient's ability to perform the exercises

Exclusion Criteria:

* severe cardiovascular disorders
* neuromusculoskeletal disorder
* cognitive impairment
* recent participation in any physiotherapy or rehabilitation program
* have exercise regularly

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
GDS-15 | 3 minutes
  consisting of 15 questions, was the primary outcome evaluator (Sheikh and Yesavage, 1986). Scores of 0-4 are considered to be normal; 5-8 indicates mild depression; 9-11 indicates moderate depression; and 12-15 indicates severe depression.
PDQ-8 | 3 minutes
  A sub-set of items is then selected from the PDQ-39 to create a shorter form version, the PDQ-8 (Jenkinson, Fitzpatrick & Peto, 1997). The sum of the scores can provide a single figure used to assess the overall health-related quality of life profile of the individual questioned. . Scores for each dimension range from 0 to 100, PDQ-8SI scores can be standardized on a scale from 0 to 100, with lower scores indicating better HRQoL.

SECONDARY OUTCOMES:
UPDRS part II (ADL) | 5 minutes
  The unified Parkinson's disease rating scale (UPDRS) is used to follow the longitudinal course of Parkinson's disease (Fahn & Elton, 1987). The UPD rating scale is the most commonly used scale in the clinical study of Parkinson's disease. A total of 199 points are possible (199 represents the worst disability and 0 no disability). Part II: self-evaluation of the activities of daily life (ADLs). The scales part 2: motor experiences of daily living (13 items), each subscale now has 0-4 ratings, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe.
UPDRS part III (motor ability) | 10 minutes
  The unified Parkinson's disease rating scale (UPDRS) is used to follow the longitudinal course of Parkinson's disease (Fahn & Elton, 1987). The UPD rating scale is the most commonly used scale in the clinical study of Parkinson's disease. Its 42 items are evaluated by interview and clinical observation. The motor section in particular to follow the progression of a person's Parkinson's disease. A total of 199 points are possible (199 represents the worst disability and 0 no disability). The scales part 3: motor examination (18 items), each subscale now has 0-4 ratings, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe.
Fatigue (FSS) | 5 minutes
  The Fatigue Severity Scale is a 9-item scale which measures the severity of fatigue (Krupp, LaRocca, Muir-Nash, & Steinberg, 1989). The subject is asked to read each statement and circle a number from 1 to 7, the items are scored on a 7 point scale with 1=strongly disagree and 7=strongly agree. The minimum score=9 and maximum score possible=63. Higher the score=greater fatigue severity.
Sleep quality (PSQI) | 5 minutes
  The Pittsburgh Sleep Quality Index (PSQI) is an effective instrument used to measure the quality and patterns of sleep in adults (Buysse, Reynolds, Monk, Berman, & Kupfer, 1989). It differentiates "poor" from "good" sleep quality by measuring seven areas (components): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction over the last month. A total score of "5" or greater is indicative of poor sleep quality.
Anxiety (HAS) | 3 minutes
  The Hospital Anxiety Scale (HAS), a self-assessment scale, was developed to detect states of, anxiety and emotional distress, used to screen for the presence of anxiety, in a general medical population of patients (Zigmond & Snaith, 1983). Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety. For both scales, scores of less than 7 indicate normal, 8-10 indicate mild anxiety, 11-14 indicate moderate anxiety and 15-21 severe anxiety.

IPD SHARING:
Plan to Share IPD: No